CLINICAL TRIAL: NCT01433055
Title: Adjunctive Minocycline in Clozapine Treated Schizophrenia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, MPRC, Deanna L. Kelly, Pharm.D., BCPP, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HP-00048900; 1R21MH091184-01A1 (NIH)
Record Dates: First submitted 2011-07-21; First posted 2011-09-13 (Estimated); Results first posted 2017-06-09 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Cognitive Symptoms; Clozapine
MeSH Terms: conditions — Schizophrenia; Neurobehavioral Manifestations | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minocycline (Active Comparator)
  Interventions: Drug: Minocycline
- Sugar Pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Minocycline — Minocycline Dosing:
  Minocycline (Dynacin® or generic) will be available in 50, 75 and 100 mg capsules. There will be matched placebo-minocycline capsules for each minocycline capsule strength. During the first week subjects will receive one 50 mg capsule twice per day (minocycline 100 mg total or matching placebo) and during weeks 2-10 subjects will receive 2- 50 mg capsules twice per day If a subject should complain of any side effect, then the blind psychiatrist will be allowed to omit the next dose of study medication and then continue the subject on the optimal treatment dose. If, despite this intervention, the subject is still unable to tolerate the 200 mg/day dose, then the dose may be lowered to 150 mg to alleviate side effects and minimize attrition.
  Arms: Minocycline
Drug: Placebo — Placebo Dosing:
  Minocycline (Dynacin® or generic) will be available in 50, 75 and 100 mg capsules. There will be matched placebo-minocycline capsules for each minocycline capsule strength. During the first week subjects will receive one 50 mg capsule twice per day(minocycline 100 mg total or matching placebo) and during weeks 2-10 subjects will receive 2- 50 mg capsules twice per day If a subject should complain of any side effect, then the blind psychiatrist will be allowed to omit the next dose of study medication and then continue the subject on the optimal treatment dose. If, despite this intervention, the subject is still unable to tolerate the 200 mg/day dose, then the dose may be lowered to 150 mg to alleviate side effects and minimize attrition.
  Arms: Sugar Pill

SUMMARY:
Schizophrenia is a devastating and costly illness. One-third to one-half of people with schizophrenia do not respond to the most current drugs leaving clozapine as the best alternative for treatment. However, over 60% of people treated with clozapine continue to have persistent symptoms and cognitive impairments. Little data is available to support evidence-based recommendations to guide clinicians in treating these patients. Preliminary data has suggested that adjunct treatment with minocycline may offer robust symptom improvement in patients with schizophrenia, including those taking clozapine. Minocycline has had interesting effects; including suggesting it may have a significant role in treatment of neurologic and psychiatric disorders. Minocycline is currently available generically; its side effects are well-described and minimal. The proposed double-blind treatment study seeks to demonstrate that adjunctive minocycline offers patients superior efficacy for persistent positive symptoms, cognitive impairments, and/or other components of schizophrenia pathology. This knowledge could lead to the more effective treatment of patients with schizophrenia. The research itself may lead to a better understanding of the pathophysiology of positive symptoms and cognitive impairments, which could contribute to improved treatments in the future.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia or schizoaffective disorder
* Male or Female
* Age: 18 to 65 years
* Caucasian or Non-Caucasian
* At least six months of clozapine treatment
* Clozapine treatment for incomplete symptoms response (evidence of two failed previous trials of antipsychotics)
* Current dose of 200 mg/day for at least 3 months AND a documented clozapine blood level 350 ng/ml prior to study start (maximum clozapine dose of 900 mg/day)
* BPRS total score of 45 or more on the 18 item version (scale: 1-7)
* BPRS positive symptom item total score of 8 or more
* BPRS positive symptom score of 4 or greater on at least one item

Exclusion Criteria:

* History of organic brain disease
* DSM-IV diagnosis of Mental Retardation
* DSM-IV diagnosis of Alcohol or Substance Dependence within the last six months (except nicotine)
* DSM-IV diagnosis of Alcohol or Substance Abuse within the last one month (except nicotine)
* Pregnancy or lactation
* Significant renal or liver impairment
* Previous known hypersensitivity to tetracyclines
* Current treatment with tetracycline or derivative
* Current treatment with lamotrigine
* Treatment with oral contraceptives
* Current known infection
* Treatment with cholestyramine or colestipol
* Treatment with Urinary alkalinizers (e.g., sodium lactate, potassium citrate)
* Treatment with warfarin
* Abnormal (considered positive) Lyme titer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deanna Kelly, Pharm.D., BCPP, Principal Investigator — University of Maryland, College Park
Locations (1):
- Maryland Psychiatric Research Center, Catonsville, Maryland, United States

REFERENCES:
- [Derived] Kelly DL, Sullivan KM, McEvoy JP, McMahon RP, Wehring HJ, Gold JM, Liu F, Warfel D, Vyas G, Richardson CM, Fischer BA, Keller WR, Koola MM, Feldman SM, Russ JC, Keefe RS, Osing J, Hubzin L, August S, Walker TM, Buchanan RW. Adjunctive Minocycline in Clozapine-Treated Schizophrenia Patients With Persistent Symptoms. J Clin Psychopharmacol. 2015 Aug;35(4):374-81. doi: 10.1097/JCP.0000000000000345. PMID 26082974

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Minocycline | Sugar Pill
Started | 29 | 23
Completed | 27 | 23
Not Completed | 2 | 0
Not completed — Diagnosed with cancer unrelated to study | 1 | 0
Not completed — Severely elevated triglycerides at entry | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minocycline | Sugar Pill | Total
Number analyzed (Participants) | 27 | 23 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (14.2) | 42.3 (11.0) | 42.6 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 19 | 18 | 37
Race/Ethnicity, Customized [Number; unit: participants]
  White | 17 | 13 | 30
  Black | 8 | 8 | 16
  Other | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 27 | 23 | 50

OUTCOME MEASURES:

1. Primary Outcome: Brief Psychiatric Rating Scale (BPRS) Positive Symptom Domain Scores Between Minocycline and Placebo.
Description: Adjunct minocycline to clozapine will be compared to placebo to test its efficacy to improve positive psychotic symptoms. The 4 item positive sub factor of the Brief Psychiatric Rating Scale (BPRS) will be the primary outcome over the 10 week randomized study. Total maximum score is 28, and total minimum score is 4. The positive domain score consists of conceptual disorganization (item 4), suspiciousness (item 11) hallucinatory behavior (item 12), and unusual thought content (item 15). All data is reported as the difference between baseline and 10 weeks. The lower the score the better the outcome.
Time Frame: 10 Weeks
Population: The BPRS is a scale that measures major psychotic and non psychotic symptoms in persons with psychotic disorders. It is an 4 item scale with a score range of 1-7 on each item. Results are reported as total score. Total maximum score is 28, and total minimum score is 4.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Minocycline | Sugar Pill
Number analyzed (Participants) | 27 | 23
units on a scale
  Baseline | 14.5 (3.5) | 14.5 (3.5)
  10 weeks (Endpoint) | 12.9 (3.2) | 14.2 (3.2)

2. Primary Outcome: Effect of Minocycline on Cognitive Symptoms as Measured by the MATRICS Consensus Cognitive Battery.
Description: Adjunct minocycline will be compared to placebo to test its efficacy in improving cognitive function. Neuropsychological testing will be done at baseline and endpoint using the MATRICS battery. A composite score as well as individual scores will be will be the primary outcome over the 10 week randomized study. This assessment total minimum score of -10 and maximum score of 80. He higher the score the better the outcome.
Time Frame: 10 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Minocycline | Sugar Pill
Number analyzed (Participants) | 27 | 23
units on a scale
  Baseline | 30.4 (11.6) | 35.1 (11.7)
  10 Weeks (Endpoint) | 35.6 (10.7) | 34.2 (12.2)

3. Secondary Outcome: The Effect of Minocycline Compared to Placebo to Improve Negative Symptoms as Measured by the Scale for the Assessment of Negative Symptoms (SANS)
Description: Adjunct minocycline will be compared to placebo to test its efficacy in improving negative symptoms of schizophrenia. The Scale for the Assessment of Negative Symptoms (SANS) will be used to test changes in the total SANS score in adjunct minocycline compared to placebo in the 10 week study. This assessment has 22 items (scored 0-5) with a total minimum score of 0 and maximum score of 110. The lower the score the better the outcome.
Time Frame: 10 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Minocycline | Sugar Pill
Number analyzed (Participants) | 27 | 23
units on a scale
  Baseline | 29.7 (13.3) | 33.3 (10.3)
  10 Weeks (Endpoint) | 28.2 (12.4) | 35.1 (10.7)

4. Secondary Outcome: The Effect of Adjunct Minocycline to Placebo to Improve Depressive Symptoms as Measured by the Calgary Depression Scale
Description: The total score of the Calgary Depression Rating Scale will be used to examine the efficacy of minocycline compared to placebo in improving depressive symptoms. This assessment has 9 items (scored 0-3) with a total minimum socre of 0 and maximum score of 27. The lower the score the better the outcome.
Time Frame: 10 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Minocycline | Sugar Pill
Number analyzed (Participants) | 27 | 23
units on a scale
  Baseline | 3.3 (3.1) | 2.6 (2.7)
  10 Weeks (Endpoint) | 2.4 (3.0) | 2.9 (2.7)

5. Secondary Outcome: The Effect of Adjunct Minocycline to Placebo on Global Clinical Improvement of Symptoms.
Description: The Clinical Global Impression Severity score will be used to examine the effect of minocycline compared to placebo. This assessment has 2 items (scored 0-7) with a total minimum socre of 0 and maximum score of 14. The lower the score the better the outcome.
Time Frame: 10 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Minocycline | Sugar Pill
Number analyzed (Participants) | 27 | 23
units on a scale
  Baseline | 4.0 (0) | 4.0 (0.1)
  10 Weeks (Endpoint) | 3.6 (0.6) | 4.0 (0.7)

ADVERSE EVENTS:
Arm/Group | Minocycline | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/23
Other Adverse Events (participants affected / at risk) | 27/27 | 22/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Minocycline (N=27) | Sugar Pill (N=23)
Nausea (Gastrointestinal disorders) | 11 | 8
Abdominal Pain (Musculoskeletal and connective tissue disorders) | 8 | 6
Vomiting (Gastrointestinal disorders) | 7 | 3
Weight loss (Metabolism and nutrition disorders) | 5 | 6
Diarrhea (Gastrointestinal disorders) | 5 | 7
Constipation (Gastrointestinal disorders) | 3 | 10
Malaise (Nervous system disorders) | 8 | 6
Sedation (Nervous system disorders) | 3 | 3
Dizziness (Nervous system disorders) | 7 | 5
Restlessness (Nervous system disorders) | 7 | 5
Salivation (General disorders) | 6 | 5
Insomnia (Nervous system disorders) | 5 | 5
Headache (General disorders) | 4 | 10
Rash (Skin and subcutaneous tissue disorders) | 4 | 1
Stiffness (Musculoskeletal and connective tissue disorders) | 4 | 5
Dry Mouth (General disorders) | 3 | 6
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No